CLINICAL TRIAL: NCT01009216
Title: A Study to Evaluate the Cerebrospinal Fluid Pharmacokinetics and Pharmacodynamics of Multiple Doses of ABT-384 in Healthy Male Volunteers
Brief Title: A Study of ABT-384 Levels and Pharmacodynamic Activity Measured in Cerebrospinal Fluid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Gerard Marek, MD, PhD, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-505
Record Dates: First submitted 2009-10-21; First posted 2009-11-06 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Pharmacology; Drug Safety; Phase 1 Clinical Trials
MeSH Terms: interventions — N-(5-(aminocarbonyl)tricyclo(3.3.1.13,7)dec-2-yl)-alpha,alpha-dimethyl-4-(5-(trifluoromethyl)-2-pyridinyl)-1-piperazineacetamide

ARMS (1):
- ABT-384 (Experimental)
  Interventions: Drug: ABT-384

INTERVENTIONS:
Drug: ABT-384 — Doses will be administered daily for 5 days.

SUMMARY:
The objectives of this study are to assess the cerebral spinal fluid (CSF) pharmacokinetics and the plasma/CSF pharmacokinetic/pharmacodynamic relationship of ABT-384 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age is between 18 and 55 years
* Judged to be in a condition of general good health based on the results of medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG

Exclusion Criteria:

* Use of protocol-prohibited medications within 2 weeks prior to study drug administration.
* Positive urine drug screen for non-prescribed drugs of abuse including alcohol.
* Receipt of any drug depot by injection within 30 days prior to study drug administration.
* Receipt of any investigational product within 6 weeks prior to study drug administration.
* History of significant sensitivity or allergy to any drug.
* History of drug or alcohol abuse.
* Positive test result for HAV, HBsAg, HCV or HIV.
* Donation or loss of 550 mL or more blood volume or receipt of any blood product within 3 months prior to study drug administration.
* Contraindication for lumbar puncture (e.g., lumbar scoliosis, coagulopathy, infected skin at puncture site)
* Current enrollment in another clinical study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability Assessments (i.e., ECG, clinical laboratory tests, vital signs, weight, AE assessment, physical and brief neurological examinations) | Days -1 through 9
Assess Pharmacokinetics (i.e., ABT-384 and possible metabolite levels) and Pharmacodynamics (i.e., biomarkers of drug effect) | Days 1, 4 through 9

CONTACTS AND LOCATIONS:
Locations (1):
- Site Reference ID/Investigator# 23882, Glendale, California, United States